CLINICAL TRIAL: NCT02375620
Title: A Multicenter, Randomized, Open-Label, Dose-Response, Phase II Clinical Study of Pegylated Somatropin (PEG Somatropin) Injection to Treat SGA Children With Short Stature.
Brief Title: Clinical Study of Pegylated Somatropin (PEG Somatropin) to Treat SGA Children With Short Stature
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Changchun GeneScience Pharmaceutical Co., Ltd. (Industry)
Collaborators: Shanxi Provincial Maternity and Children's Hospital (Other); Children's Hospital of Fudan University (Other); Xinhua Hospital, Shanghai Jiao Tong University School of Medicine (Other); The First Hospital of Jilin University (Other); Hunan Children's Hospital (Other Government); Tongji Hospital (Other); Affiliated Hospital of Jiangnan University (Other); Jiangxi Province Children's Hospital (Other); Children's Hospital of The Capital Institute of Pediatrics (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GenSci 031 CT
Record Dates: First submitted 2015-02-01; First posted 2015-03-02 (Estimated); Last update posted 2025-05-25 (Actual); Status verified 2025-05

CONDITIONS: Short Stature Children Born Small for Gestational Age (SGA)

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- PEG-somatropin: Low dose (Experimental): 0.1 mg/(kg.w), once per week for 52 weeks.
  Interventions: Biological: PEG-somatropin
- PEG-somatropin: High dose (Experimental): 0.2 mg/(kg.w), once per week for 52 weeks.
  Interventions: Biological: PEG-somatropin
- Children who completed the 52- week main phase proceeded to the extension phase (Experimental): Dose adjustments based on annualized height velocity (AHV; cm/year) and insulin-like growth factor I (IGF-I) response, were made up to a maximum of 0.4 mg/kg/week until achieved NAH or the patient's voluntary discontinuation.
  Interventions: Biological: PEG-somatropin

INTERVENTIONS:
Biological: PEG-somatropin

SUMMARY:
The study was evaluated as the optimal dose for the treatment of SGA short stature children by Pegylated Somatropin, initially evaluated its efficiency and safety for the treatment of SGA short stature children and provided scientific, reliable basis for phase III clinical trials for dose selection.

This is a multicenter, randomized, open-label, dose-response trial, including a 52-week main phase and an ongoing safety extension phase continuing until reaching near-adult height (NAH) in China. Ninety-six growth hormone (GH)-treatment-naïve, non-GH-deficient, prepubertal short children born SGA were randomized in a 1:1 ration to receive weekly subcutaneous administration of Jintrolong 0.1 mg/kg/week or 0.2 mg/kg/week for 52 weeks. Children who completed the 52- week main phase proceeded to the extension phase, while Jintrolong was administered at an initial dose of 0.2 mg/kg/week. Dose adjustments based on annualized height velocity (AHV) and insulin-like growth factor I (IGF-I) response, were made up to a maximum of 0.4 mg/kg/week until achieved NAH or the patient's voluntary discontinuation.

ELIGIBILITY:
Inclusion Criteria:

* The patients are diagnosed as being clinically full term small for gestational age infant.
* Girl are 3-6 years old, boys are 3-7 years old.
* Be in preadolescence (Tanner stage 1).
* The child did not achieve catch-up growth when he/she entered the group (the definition of catch-up growth is that the height is higher the third percentile with the same age and gender) (Appendix 2 and 3).
* The height of child is shorter than -2SDS of the median of normal children with the same age and gender when he/she entered the group (the mean height and height standard deviation of normal children with the same age and gender of normal children regard the height data in the physical development investigation data of children aged 0-18 in 9 cities of China (2005) as standard [13], Appendix 4 and 5).
* Within a year before entering the group, after any growth hormone stimulation test, the peak concentration of growth hormone in serum>10 µg/L.
* Bone age≤ the actual age+1.
* The function of glucose regulation is normal: fasting blood glucose < 5.6mmol/L.
* Birth gestational age ≥ 37 weeks.
* The subjects and their guardians sign the informed consent (if the subjects is lack of ability for signing the informed consent, his legal guardian can write the subjects name instead).
* All experimental drug groups completed the main phase (52 weeks) of Phase II clinical trials, and the participants with complete follow-up records can enter the extension phase, provided that the continuous cessation of the use of pegylated recombinant human growth hormone injection lasts ≤ 8 weeks after the end of the first phase treatment and before the start of the extended study.
* Only when the subjects and their guardians are fully informed, express their willingness, and are able to cooperate in completing the treatment, follow-up, and various tests of the extension phase study, and have signed a written informed consent form, can they enter the extension phase trial.

Exclusion Criteria:

* People with abnormal liver or kidney function (ALT> 2 times the upper limit of normal value, Cr> the upper limit of normal value).
* Patients are positive for hepatitis B core antigen (HBc), hepatitis B surface antigen (HBsAg) or hepatitis B e antigen (HBeAg).
* People with known highly allergic constitution or allergy to the drug or the excipient of the study.
* People with diabetes, severe cardiopulmonary, hematological system and malignant tumors diseases or general infection, immune deficiency and patients with mental disease.
* Other abnormal growth and development, such as Turner syndrome, Laron syndrome, growth hormone receptor deficiency.
* Potential tumor patients (family history).
* Patients who used growth hormone for treatment.
* Subjects took part in other clinical trial study within 3 months.
* Patients used other hormonal for treatment within 3 months (such as sex hormone, glucocorticoid and etc., treat for more than a month) and received the drug treatment which may interfere with the secretion of GH or GH function (oxandrolone, growth hormone releasing hormone and etc.);
* Other conditions which in the opinion of the investigator preclude enrollment into the study.
* Subjects who have used the following medications within 2 months prior to entering the expansion phase of the trial:
* 1) Aromatase inhibitors (including but not limited to letrozole, anastrozole) used continuously for 1 month;
* 2) Gonadotropin-releasing hormone analogs (including but not limited to triptorelin, leuprolide, goserelin) used continuously for 1 month;
* 3) Sex hormones (including but not limited to any type of estrogen, progestin, and androgen) used continuously for 1 month;
* 4) Anabolic steroids (including but not limited to oxymetholone, danazol, stanozolol) used continuously for ≥ 1 month;
* 5) Oral or intravenous corticosteroids used for 1 month.

Ages: 3 Years to 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 96 (Estimated)
Dates: Start 2015-04-23 (Actual); Primary Completion 2023-12-12 (Actual); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
The change in height standard deviation scores (HT SDS) of the chronological age from baseline. | The main phase is at 52 weeks and the extension phase is at every 52 weeks up to study completion.

SECONDARY OUTCOMES:
Annualized Height Velocity | The main phase is at 52 weeks and the extension phase is at every 52 weeks up to study completion.
The change of height from baseline | The main phase is at 52 weeks and the extension phase is at every 52 weeks up to study completion.
Bone maturity (bone age/ chronological age , △BA/△CA ) | The main phase is at 52 weeks and the extension phase is at every 52 weeks up to study completion.
The change of IGF-1 standard deviation scores(IGF-1 SDS) from baseline | The main phase is at 52 weeks and the extension phase is at every 52 weeks up to study completion.
The change of mole ratio of IGF-1/IGFBP-3 from baseline | The main phase is at 52 weeks and the extension phase is at every 52 weeks up to study completion.
The change of BMI standard deviation scores(BMI SDS) | The main phase is at 52 weeks and the extension phase is at every 52 weeks up to study completion.

CONTACTS AND LOCATIONS:
Overall Officials: Xiaoping Luo, Ph.D, Principal Investigator — Tongji Hospital
Locations (9):
- China (9):
  - Children's Hospital, Capital Institute of Pediatrics, Beijing, Beijing Municipality
  - Tongji Hospital, Tongji Medical College, Huazhong University of Science & Technology, Wuhan, Hubei
  - Hunan Children's Hospital, Changsha, Hunan
  - Affiliated Hospital of Jiangnan University, Wuxi, Jiangsu
  - Jiangxi Provincial Children's Hospital, Nanchang, Jiangxi
  - First Hospital of Jilin University, Changchun, Jilin
  - Children's Hospital of Fudan University, Shanghai, Shanghai Municipality
  - Xinhua Hospital Affiliated to Shanghai Jiaotong University School of Medicine, Shanghai, Shanghai Municipality
  - Shanxi Children's Hospital/Shanxi Women and Children Hospital, Taiyuan, Shanxi

REFERENCES:
- [Derived] Luo X, Hou L, Zhong Y, Zhao S, Chen X, Dong Q, Du H, Lu H, Yang Y, Wu X, Luo F, Chen R, Xu Z, Ma Y, Song W, Feng M, Gu X, Qiu W. A Phase 2 Study of PEGylated Recombinant Human Growth Hormone for 52 Weeks in Short Children Born Small for Gestational Age in China. Clin Endocrinol (Oxf). 2025 Feb;102(2):136-146. doi: 10.1111/cen.15156. Epub 2024 Nov 8. PMID 39513569